CLINICAL TRIAL: NCT05398783
Title: A Natural History Study of Metabolic Sizing in Health and Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000617; 000617-DK
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12-23

CONDITIONS: Metabolic Disorders; Cancer; Chronic Kidney Disease; Diabetes; Normal Physiology
Keywords: Body Composition; Metabolism; Body Surface Area; Natural History
MeSH Terms: conditions — Metabolic Diseases; Neoplasms; Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Male and female volunteers aged 2+ years in good general health as evidenced by medical history
- Patients: Male and female patients aged 2+ years diagnosed with diseases thought to alter metabolism or body composition and/or taking medication thought to alter metabolism or body composition

SUMMARY:
Background:

Scientists have long used simple measures (such as height and weight) to estimate how much a person s body uses food (calories) as energy, as commonly called the metabolic rate. But metabolism varies among people with similar body sizes. Scientists now believe the old formulas for estimating metabolic rates may not work well for all people. Researchers want to find more accurate ways to measure a person s metabolism.

Objective:

This natural history study will examine the relationships between metabolism, body composition, and body surface area in a wide range of people.

Eligibility:

Healthy children and adults aged 2 years or older. Also, people aged 2 years or older with conditions that may alter metabolism. These may include diabetes, obesity, renal disease, or cancer.

Design:

Participants will spend 2 days and 1 night in the hospital. They will provide a medical history and answer questions about their activity levels, the foods they eat, and their lifestyle. They will also eat a special diet.

Participants will undergo many tests:

They will lie in a bed with a clear hood covering their head for 30 to 45 minutes to measure the gases in their breath.

They will lie on a padded table for about 15 minutes while their body is scanned.

They will stand on a platform while a 3D scanner measures their body.

They will have a test to measure how fast an electric signal moves through their body.

They will grip an instrument to measure the strength of their hands.

They will drink salty water and provide blood and urine samples.

Participants may be invited to return for these 2-day visits up to 8 times per year. Return visits must be at least 2 weeks apart.

DETAILED DESCRIPTION:
Study Description:

This study will examine the relationships between comprehensively measured resting energy expenditure (REE), body composition, and body surface area (BSA) in a wide range of healthy and diseased individuals.

Objectives:

Primary Objectives:

* To compare estimated and measured BSA.
* To determine if measured BSA is associated with REE independent of body composition measures

Endpoints:

Primary Endpoints:

* Mean difference and limits of agreement at baseline between measured BSA and predicted BSA calculated from traditional biometrics such as height and weight.
* Increase in R^2 when measured BSA is added to equations predicting REE.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all the following criteria for their cohort:

Cohort 1 - Healthy Volunteers

* Male or female, aged >=2 years
* In good general health as evidenced by medical history

Cohort 2 - Patients

* Male or female, aged >=2 years
* Diagnosed with diseases thought to alter metabolism or body composition (such as weight loss or gain, diabetes, renal disease, obesity, cancer, etc.) or taking medications thought to alter metabolism or body composition.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Participants over 200 kg due to the weight limit of the equipment.
* Presence of any implanted device that would interfere with measurements.
* Any moderate to severe limitations in mobility that would impede participation
* Hemoglobin less than 10 g/dL (in participants who would have blood drawn for research purposes)
* Participants with dietary allergies, intolerances or eating patterns that would preclude them from consuming metabolic meals.
* Participants unwilling or unable to give informed consent.
* Participants with any other significant physical, medical, or psychiatric limitations, illness or conditions that may preclude them from completing the majority of the tests in this study per the discretion of the PI.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Local population, primary clinical, referred patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Increase in R^2 | Per study visit
  Increase in R2 when measured BSA is added to equations predicting REE
Mean difference and limits of agreement between measured and predicted BSA | Per study visit
  Mean difference and limits of agreement between measured BSA and predicted BSA calculated from traditional biometrics such as height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ishihara A, Brychta RJ, LaMunion SR, McGehee S, Donayre M, Jordan O, Davis K, Sanchez G, Smith L, Chung ST, Courville AB, Chen KY. Performance of wearable light sensors for measuring photopic and melanopic illuminance under laboratory and free-living conditions. Sleep. 2026 Feb 10;49(2):zsaf358. doi: 10.1093/sleep/zsaf358. PMID 41230818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000617-DK.html